CLINICAL TRIAL: NCT03063827
Title: Effect of Botulinum Toxin A on Neurogenic Detrusor Overactivity in Chronic Spinal Cord Injured Patients - An Investigation of Sensory Receptor Expressionsbetween Responders and Non-responders
Brief Title: Effect of Botulinum Toxin A on Neurogenic Detrusor Overactivity in Chronic Spinal Cord Injured Patients
Status: Completed | Type: Observational
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Chairman, Department of Urology, Buddhist Tzu Chi General Hospital
Other Study IDs: BuddhistTCGH 098-53
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Neurogenic Bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment group: Patients with chronic SCI causing NDO and urinary incontinence
  Interventions: Drug: OnabotulinumtoxinA 200 UNT; Diagnostic Test: Urothelial sensory protein levels
- Control group: Female patients who underwent anti-incontinence suregery without lower urinary tract symptoms
  Interventions: Diagnostic Test: Urothelial sensory protein levels

INTERVENTIONS:
Drug: OnabotulinumtoxinA 200 UNT — Patient in the treatment arm received a single injection of onabotulinumtoxinA 200 UNT to the detrusor muscle at 20 sites of the bladder body.
  Other Names: OnabotulinumtoxinA (Botox) 200 UNT
  Groups: Treatment group
Diagnostic Test: Urothelial sensory protein levels — Bladder tissues were investigated for urothelial barrier and inflammation proteins as well as urothelial sensory protein levels by Western blotting, between SCI patients and 10 controls, as well as successful and failed treatment groups.
  Other Names: Sensory proteins

SUMMARY:
This study investigated the changes in urothelial dysfunction and sensory protein expression in the bladder urothelium with time after onabotulinumtoxin injection in spinal cord injured (SCI) patients. The investigators planned to enroll 30 chronic SCI patient with neurogenic detrusor overactivity and urinary incontinence were treated with a single injection of 200 U onabotulinumtoxinA at the detrusor. Video urodynamic studies and bladder mucosal biopsies were performed at baseline, 3 months, and 6 months after treatment. Bladder tissues will be investigated for urothelial barrier and inflammation proteins as well as sensory proteins by Western blotting, between SCI patients and 10 controls, as well as successful and failed treatment groups. This study will explore the therapeutic efficacy of a single injection of 200 U onabotulinumtoxinA on neurogenic detrusor overactivity and the changes of urothelial sensory proteins in SCI patients with successful and failed treatment outcome.

DETAILED DESCRIPTION:
In recent decades, treatment of neurogenic detrusor overactivity (NDO) with onabotulinumtoxinA has emerged as an alternative method for the management of urological complications due to spinal cord injury (SCI) or multiple sclerosis. Injection of 200-300 U of onabotulinumtoxinA into the detrusor muscle can reduce contractility, improve bladder compliance, and restore urinary continence in patients with NDO. However, detrusor underactivity will develop after injection of 300 U of onabotulinumtoxinA and improvement of urodynamic and quality of life parameters lasted 9 months. Currently, a 200 U single injection of onabotulinumtoxinA into the detrusor has been recommended as standard treatment for NDO. However, the therapeutic duration of this dosage on NDO was shorter than that of a 300 U injection.

OnabotulinumtoxinA effectively improves lower urinary tract symptoms by inhibiting signal transmission at the neuromuscular and neuroglandular junctions. OnabotulinumtoxinA cleaves synaptosome-associated protein 25 and inhibits signal transmission by disrupting fusion of neurotransmitter- containing vesicles with the neuronal wall. In the urinary bladder, release of acetylcholine from both pre- and postganglionic parasympathetic nerves is blocked after onabotulinumtoxinA administration. This toxin was also found to modulate afferent activity of the bladder associated with reduced urgency and urgency urinary incontinence symptoms in NDO patients. Although the impact of onabotulinumtoxinA on the sympathetic nervous system within the urinary bladder is unclear, it has an inhibitory effect on release of norepinephrine to α- and β3-adrenoreceptors (β3-ARs) which regulate bladder neck contraction and detrusor relaxation, respectively.

A previous study reported decreased expression of adhesion and junction proteins E-cadherin and zonula occludens-1 (ZO-1), respectively, and increased suburothelial inflammation with apoptosis in patients with chronic SCI bladders.The urothelial inflammation and dysfunction in SCI bladders might also alter sensory protein expression, such as in purinergic receptor P2X3, transient receptor potential vallinoid receptor subfamily 1, adenosine triphosphate, and nitric oxide. Urothelial dysfunction might also result in increased excitability of the C-fibers which become predominantly afferent nerves of the micturition reflex after SCI. In humans with NDO, the levels of bladder P2X2, P2X3, and muscarinic receptors M2 and M3 were reduced after detrusor onabotulinumtoxinA injection, suggesting this toxin inhibits DO by inhibiting both the sensory and motor arms of the micturition reflex. In addition, β3-ARs are known to promote urine storage in the bladder by inducing detrusor relaxation in animal and human bladders. In humans, β3-AR is the predominant β-receptor subtype in the urinary bladder. There has been no report on β3-AR changes in SCI bladder urothelium before or after onabotulinumtoxin treatment.

After onabotulinumtoxinA injection, patients may be symptom-free for a period of 3-6 months before symptoms relapse. Most studies of onabotulinumtoxinA on NDO come from animal models, and only a few human studies have been noted. The current study investigated changes in urothelial dysfunction and sensory protein expression in the bladder urothelium with time after a single onabotulinumtoxin injection in SCI patients.

Materials and Methods

A total of 26 patients with chronic SCI causing NDO and urinary incontinence were treated with a single injection of 200 U onabotulinumtoxinA to the detrusor muscle. All patients presented with urinary incontinence with or without difficult bladder emptying. In patients who received detrusor injections, clean intermittent catheterization was suggested as a possible mode of urinary management after treatment. The current study was approved by the Institutional Review Board and Ethics Committee of Buddhist Tzu Chi General Hospital (IRB:098-53). Each patient was informed about the study rationale and procedures, and written informed consent to participate was obtained before any bladder procedure.

Video urodynamic studies

All patients received a video urodynamic study (VUDS) before their enrollment. Bladder and urethral dysfunction were classified as the presence of DO with coordinated or dyssynergic urethral sphincter activity. Patients with urinary tract infection were properly treated before they were scheduled for onabotulinumtoxinA injection. VUDS results were interpreted according to the recommendations of the International Continence Society. VUDS parameters included maximum flow rate (Qmax), detrusor voiding pressure at Qmax (Pdet), cystometric bladder capacity (CBC), voided volume (Vol), and post-void residual (PVR) volume.

OnabotulinumtoxinA injection

All patients received 200 U of onabotulinumtoxinA in 20 mL normal saline (BOTOX®, 100 U/vial, Allergan Inc., Irvine, USA) in the operation room by rigid cytoscopic injection (22 Fr, Richard Wolf, Knittlingen, Germany) into 40 sites of the bladder wall, sparing the trigoneAfter injection, a urethral Foley catheter was routinely inserted and removed the next morning before patients were discharged. Broad spectrum antibiotics were prescribed for 3 d after treatment.

After onabotulinumtoxinA injection, four bladder cold-cup biopsies were taken randomly at the posterior wall about 2 cm above the interureteric ridge, and only the bladder mucosa and submucosa were taken to prevent bladder perforation; any erythematous or inflammatory bladder mucosa were avoided. One bladder biopsy specimen from each patient was sent to the pathology department to exclude the possibility of carcinoma in situ. The remaining three specimens from each patient were stored at optimum cutting temperature and in liquid nitrogen for further immunohistochemistry studies.

Patient follow-up and outcome assessment

Patients were followed up at OPD monthly, and VUDS and assessment of bladder and voiding conditions and satisfaction with treatment were performed 3 and 6 months after treatment. If the CBC increased by 50% from the baseline value, the treatment outcome was considered successful; otherwise, the outcome was considered a failure at that time-point. Ten female patients with stress-related urinary incontinence without frequent urgency served as controls. All control patients were confirmed free of bladder outlet obstruction or DO by VUDS. Control bladder tissue was obtained during anti-incontinence surgery and processed the same as SCI patients. Male patients were not selected to serve as controls because the prostate could cause bladder outlet obstruction and affect urothelial function.

Immunofluorescence

Bladder tissue samples from SCI patients and controls were examined for changes in urothelial E-cadherin (adhesive protein), ZO-1 (junction protein), and mast cell activation (tryptase) levels by immunofluorescence; cellular apoptosis was examined by terminal deoxynucleotidyl transferase dUTP nick end-labeling assay. These procedures were performed similar to those in our previous study, with 6-μm thickness tissue sections. Urinary bladder specimens were immersed and fixed for 1 h in ice-cold 4% formaldehyde in phosphate-buffered saline (pH 7.4) then rinsed with ice-cold phosphate-buffered saline containing 15% sucrose for 12 h. Biopsy specimens were embedded in optimum cutting temperature medium and stored at -80 °C. Four sections per specimen were cut using a cryostat at a thickness of 8 μm and collected on new silane III-coated glass slides (Muto Pure Chemicals Co., Ltd, Tokyo, Japan). Sections were postfixed in acetone at -20 °C and blocked with rabbit serum. The sections were incubated overnight at 4 °C with antihuman E-cadherin (BD Biosciences, San Jose, CA, USA) or tryptase (Chemicon, Temecula, CA, USA) primary antibodies. After rinsing the sections with 0.1% Tween-20 in BPS, rabbit antimouse-conjugated fluorescein isothiocyanate secondary antibodies (DakoCytomation Denmark A/S, Glostrup, Denmark) were applied and incubated on sections for 1 h. Finally, sections were counterstained with 4',6-diamidino-2-phenylindole (Sigma Chemical Co., St. Louis, MO, USA). Negative controls included the isotype of the primary antibody. We obtained the mean, maximum, range, and standard deviation of the staining intensity and percent positive area measurements using three random hot spots within each specimen.

Immunofluorescence quantification was determined in four consecutive high-power fields (400X) in the area with the greatest density. Immunofluorescence (tryptase and terminal deoxynucleotidyl transferase dUTP nick end-labeling) assays were quantified by counting the number of positively stained cells per unit area (4 μm2) and are shown as percentages. The intensity of E-cadherin (ﬂuorescence microscopy) and ZO-1 (confocal microscopy) fluorescence was quantified using Image J.

Western blotting was used to assess the levels of sensory proteins in bladder mucosa specimens. Primary antibodies included P2X3 (1:2000), endothelial nitric oxide synthase [eNOS] (1:1000), M2 (1:1000), M3 (1:500), and GAPDH (1:100000; internal control) from GeneTex (Irvine, CA, USA); inducible NOS [iNOS] (1:1500; ThermoFisher, Rockford, IL, USA); and β3-AR (1:1000; Abcam, Cambridge, UK). Donkey antigoat (for β3-AR) or goat antirabbit (for all other proteins) IgG-horseradish peroxidase (1:3000; Santa Cruz Biotechnology, Dallas, TX, USA) secondary antibodies were used. The scanned ﬁlm after gel electrophoresis was quantiﬁed using a gel documentation system (Quantity One Version 4.6.2, Bio-Rad Laboratories, Hemel Hempstead, Herts, UK). Procedures were similar to those described in our previous study.

Statistical Analysis

Continuous variables were presented as means ± standard deviations, and categorical data were presented as numbers and percentages. Eligible SCI patients were grouped according to treatment outcome and compared with controls. Differences in the levels of functional proteins in the urothelium at baseline and 3 and 6 months after onabotulinumtoxinA injection were analyzed using a paired Student's t-test. Differences in immunofluorescence and Western blot of sensory proteins between successful and failed treatment groups were analyzed using the Kruskal-Wallis test. In order to clarify the roles of urothelial sensory proteins in NDO, correlation analysis using linear regression was also performed, including VUDS and urothelial dysfunction parameters. All calculations were done using SPSS for Windows version 16.0 (SPSS, Chicago, IL, USA). Differences were considered statistically significant if P values were less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic SCI causing NDO and urinary incontinence

Exclusion Criteria:

* patients did not present with urinary incontinence
* patients are known to be allergic to onabotulinumtoxinA
* patients cannot be followed up regularly
* active urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with chronic spinal cord injury causing neurogenic detrusor overactivity and urinary incontinence were treated with a single injection of 200 U onabotulinumtoxinA to the detrusor muscle. All patients presented with urinary incontinence with or without difficult bladder emptying. In patients who received detrusor injections, clean intermittent catheterization was suggested as a possible mode of urinary management after treatment.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Bladder capacity | from baseline to 6 months after treatment
  The maximal cystometric or functional bladder capacity

SECONDARY OUTCOMES:
IIQ-7 | from baseline to 6 months after treatment
  Incontinence impact questionnare score
UDI-6 | from baseline to 6 months after treatment
  Urogenital distress inventory score
Sensory protein assessment | from baseline to 6 months after treatment
  The changes of urothelial sensory protein levels

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to share with other researchers